CLINICAL TRIAL: NCT01426490
Title: The Effects of Vitamin B-6 Status on Homocysteine, Oxidative Stress, One-carbon Metabolism and Methylation: Cross-section, Case-control, Intervention and Follow-up Studies in Colorectal Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: S10251
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2011-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ascorbic Acid; Vitamin B 6; Pyridoxine; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin C (Other): Vitamin C as control group.
  Interventions: Dietary Supplement: Vitamin C
- Vitamin B6 (Experimental)
  Interventions: Dietary Supplement: Vitamin B6
- Folic acid (Experimental)
  Interventions: Dietary Supplement: Folic acid
- Vitamin B6 plus folic acid (Experimental)
  Interventions: Dietary Supplement: Vitamin B6 plus folic acid

INTERVENTIONS:
Dietary Supplement: Vitamin C — Vitamin C, 100 mg/d
  Other Names: Ascorbic acid
  Arms: Vitamin C
Dietary Supplement: Vitamin B6 — Vitamin B6, 50mg/d
  Other Names: Pyridoxine
  Arms: Vitamin B6
Dietary Supplement: Folic acid — Folic acid 400 microgram/d
  Other Names: Folate
  Arms: Folic acid
Dietary Supplement: Vitamin B6 plus folic acid — Vitamin B6, 50 mg; folic acid, 400 microgram
  Other Names: B-vitamins (pyridoxine and folate)
  Arms: Vitamin B6 plus folic acid

SUMMARY:
Vitamin B-6, folate and homocysteine may play a critical role in the colorectal cancer progression. This is a 4-y study and the specific aims are: 1) to compare vitamin B-6, folate and homocysteine status, oxidative stress, antioxidant activities and DNA methylation between subjects with colorectal polyps and colorectal cancer; 2) to study the effects of vitamin B-6, folate and homocysteine status on oxidative stress, antioxidant activities and DNA methylation in colorectal cancer patients; 3) to evaluate whether folic acid and/or pyridoxine supplementation had a beneficial effect on oxidative stress, antioxidant activities and DNA methylation in patients with colorectal; 4) to compare vitamin B-6, folate and homocysteine status, oxidative stress, antioxidant activities and DNA methylation between colorectal cancer patients and age-, sex-matched healthy subjects; 5) to evaluate the effect of vitamin B-6, folate and homocysteine status, oxidative stress, antioxidant activities and DNA methylation on the risk of colorectal cancer (odds ratio); 6) to follow the effects of vitamin B-6, folate and homocysteine status, oxidative stress, antioxidant activities and DNA methylation on the occurrence of colorectal cancer; 7) to follow the effects of pyridoxine and/or folic acid supplementation on the occurrence of colorectal cancer.

This protocol is designed as a hospital-based cross-sectional, case-control, double blinded randomized placebo-controlled intervention and follow-up trial. Three hundred colorectal cancer patients and 300 age-, sex-matched controls who meet the inclusion criteria will be recruited from Taichung General Veterans Hospital. If cancer patients' plasma pyridoxal 5'-phosphate (PLP) level less than 30 nmol/L will be asked to participate the intervention study and will be blinded and randomly assigned to either the 1) control (vitamin C, 100 mg/d); 2) 50 mg vitamin B-6; 3) 400 microgram/d folic acid; or 4) vitamin B-6 (50 mg/d) plus folic acid (400 microgram/d) for 1 year. Data on demography, anthropometry, medical history, food frequency questionnaire and 24-h diet recall will be collected. Cancer patients will have fasting blood drawn before surgery or receiving chemotherapy. Additionally, fasting blood samples will be obtained at month 0, 3, 6, 9 and 12 during intervention period and at month 6, 12, 18, 24, 30, 36, 42 and 48 during follow-up. Hematological, plasma and erythrocyte PLP, plasma pyridoxal and 4-pyridoxic acid, serum and erythrocyte folate, serum vitamin B-12, homocysteine, SAM, SAH, lipid peroxidation indicators (TBARS, oxidized LDL), glutathione, antioxidant enzymatic activities and DNA methylation and MTHFR 677C>T polymorphism will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer participants were identified by colonoscopy to have at least one historically confirmed colorectal cancer.

Exclusion Criteria:

* Age<18 years
* Pregnant women
* Had a history of colorectal cancer
* Attenuated adenomatous polyposis coli
* Inflammatory bowel disease or were taking any medication which could influence homocysteine, folate, vitamin B6 and B12 status, such as H2 blockers, Proton pump inhibitors, metformin, phenytoin, methotrexates.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Antioxidant and DNA methylation | 12 months
  This study are going to measure the oxidative stress (TBARs), antioxidant activities and DNA methylation in colorectal cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Verterans General Hospital, Taichung, Taiwan